CLINICAL TRIAL: NCT01430611
Title: Safety and Immunogenicity of Sanofi Pasteur Meningococcal (Groups A and C) Polysaccharide Vaccine Versus Lanzhou Institute for Biological Products Meningococcal (Groups A and C) Polysaccharide Vaccine in Children 2-6 Years of Age in China
Brief Title: Study of Sanofi Pasteur and Lanzhou Institute's Meningococcal (Group A and C) Polysaccharide Vaccine in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MPS01; U1111-1120-1190 (Other: WHO)
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Meningococcal Disease; Meningitis
Keywords: Meningitis; Neisseria meningitidis; Meningo A+C®; Meng Ling Kang®
MeSH Terms: conditions — Meningococcal Infections; Meningitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine (Experimental)
  Interventions: Biological: Meningococcal (Groups A and C) Polysaccharide Vaccine
- Lanzhou Institute Meningococcal A+C Polysaccharide Vaccine (Active Comparator)
  Interventions: Biological: Meningococcal (Groups A and C) Polysaccharide Vaccine

INTERVENTIONS:
Biological: Meningococcal (Groups A and C) Polysaccharide Vaccine — 0.5 mL, Subcutaneous
  Other Names: Meningo A+C®
  Arms: Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine
Biological: Meningococcal (Groups A and C) Polysaccharide Vaccine — 0.5 mL, Subcutaneous
  Other Names: Meng Ling Kang®
  Arms: Lanzhou Institute Meningococcal A+C Polysaccharide Vaccine

SUMMARY:
This study is part of the post-licensure commitment to evaluate the safety and immunogenicity of Meningo A+C vaccine in healthy Chinese children 2 to 6 years of age.

Primary Objective:

To demonstrate the non-inferiority in terms of seroconversion rate for serogroups A and C, 30 days after a single dose of Sanofi Pasteur Meningococcal (Groups A and C) Polysaccharide Vaccine versus Lanzhou Institute for Biological Products Meningococcal (Groups A and C) Polysaccharide Vaccine.

Secondary Objective:

* To describe the immunogenicity for serogroups A and C, 30 days after administration of the study vaccines given as a single dose.
* To describe the full reactogenicity profile after administration of the study vaccines given as a single dose.

DETAILED DESCRIPTION:
Eligible participants will receive one injection of either Sanofi Pasteur Meningococcal (Groups A and C) Polysaccharide Vaccine or Lanzhou Institute for Biological Products Meningococcal (Groups A and C) Polysaccharide Vaccine and will be monitored for safety and immunogenicity for up to 30 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 6 years on the day of inclusion
* Informed consent form has been signed and dated by the parent or another legally acceptable representative
* Subject and parent/ legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures
* Written documentation of immunization history against meningococcal disease according to the national Expanded Program on Immunization (EPI) schedule (including 2 doses with Meningococcal Group A Polysaccharide Vaccine between 6 and 18 months of age).

Exclusion Criteria:

* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following the trial vaccination (except for influenza vaccination, which may be received at least 2 weeks before study vaccines)
* Previous vaccination against meningococcal disease within the past 12 months with either the trial vaccine or another vaccine
* Previous vaccination with any meningococcal conjugate vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically
* At high risk for meningococcal disease during the trial, including:

  1. persons with increased susceptibility such as persistent complement component deficiencies,
  2. persons with anatomic or functional asplenia,
  3. persons who have exposure (e.g., microbiologists routinely working with N. meningitidis, or travelers to or residents of areas where meningococcal disease is hyperendemic or epidemic)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Known thrombocytopenia, as reported by the parent/ legally acceptable representative, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥ 37.1°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of oral or injected antibiotic therapy within 72 hours before the first blood draw
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study
* Any contraindication as listed in the study vaccines leaflets.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 666 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (2):
- China (2):
  - Chuzhou
  - Nanjing

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 23 August 2011 to 12 October 2011 at a single center in China.
Pre-assignment Details: A total of 665 of the 666 participants who met all of the inclusion and none of the exclusion criteria that were randomized were vaccinated in this study.
Groups:
- Meningo A+C® (Group 1): Children aged 2 to 6 years received a single dose of Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine
- Meng Ling Kang® (Group 2): Children aged 2 to 6 years received a single dose of Lanzhou Institute of Biological Products Meningococcal A+C Polysaccharide Vaccine
Period: Overall Study
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2)
Started | 332 | 333
Completed | 315 | 318
Not Completed | 17 | 15
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2) | Total
Number analyzed (Participants) | 332 | 333 | 665
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 332 | 333 | 665
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.2 (1.1) | 3.1 (1.0) | 3.2 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 133 | 277
  Male | 188 | 200 | 388
Region of Enrollment [Number; unit: Participants]
  China | 332 | 333 | 665

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroconversion Following Vaccination With Either Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine or Lanzhou Institute of Biological Products Meningococcal A+C Polysaccharide Vaccine
Description: Seroconversion status was defined as antibody titers against meningococcal serogroups A and C, 30 days after vaccine administration ≥ 4-fold increase from pre-vaccination level measured by 2,3,5 triphenyltetrazolium chloride (TTC) serum bactericidal assay using baby rabbit complement (SBA-BR).
Time Frame: Day 30 post-vaccination
Population: Seroconversion was assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2)
Number analyzed (Participants) | 304 | 308
Participants
  Serogroup A (N = 304, 308) | 295 | 301 [0 to 0]
  Serogroup C (N = 304, 308) | 288 | 292 [0 to 0]

2. Secondary Outcome: Percentage of Participants With Post-vaccination Titer ≥1:8 for Serogroup A Before and Following Vaccination of Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine or Lanzhou Institute of Biological Products Meningococcal A+C Polysaccharide Vaccine
Description: Meningococcal Group A antibodies were measured by 2,3,5 triphenyltetrazolium chloride (TTC) serum bactericidal assay using baby rabbit complement (SBA-BR)..
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Immunogenicity was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2)
Number analyzed (Participants) | 304 | 308
Percentage of participants
  Serogroup A (pre-vaccination) | 12.5 | 8.8 [0 to 0]
  Serogroup A (post-vaccination) | 98.0 | 99.0 [0 to 0]

3. Secondary Outcome: Percentage of Participants With Post-vaccination Titer ≥1:8 for Serogroup C Before and Following Vaccination of Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine or Lanzhou Institute of Biological Products Meningococcal A+C Polysaccharide Vaccine
Description: Meningococcal Group C antibodies were measured by 2,3,5 triphenyltetrazolium chloride (TTC) serum bactericidal assay using baby rabbit complement (SBA-BR)..
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Immunogenicity was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2)
Number analyzed (Participants) | 304 | 308
Percentage of participants
  Serogroup C (pre-vaccination) | 25.0 | 26.0 [0 to 0]
  Serogroup C (post-vaccination) | 97.0 | 96.8 [0 to 0]

4. Secondary Outcome: Geometric Mean Titers of Serogroup A and C Antibodies Following Vaccination With Either Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine or Lanzhou Institute of Biological Products Meningococcal A+C Polysaccharide Vaccine
Description: Meningococcal Group A and C antibodies were measured by 2,3,5 triphenyltetrazolium chloride (TTC) serum bactericidal assay using baby rabbit complement (SBA-BR).
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Geometric mean titers were assessed in the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2)
Number analyzed (Participants) | 332 | 333
Titers
  Serogroup A (pre-vaccination; N = 332, 333) | 1.75 [1.52 to 2.00] | 1.45 [1.29 to 1.63]
  Serogroup A (post-vaccination; N = 315, 318) | 207 [182 to 236] | 223 [201 to 248]
  Serogroup C (pre-vaccination; N = 332, 333) | 3.57 [3.20 to 3.97] | 3.65 [3.28 to 4.07]
  Serogroup C (post-vaccination; N = 315, 318) | 181 [158 to 208] | 192 [168 to 220]

5. Secondary Outcome: Geometric Mean Titers of Serogroup A Antibodies Following Vaccination With Either Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine or Lanzhou Institute of Biological Products Meningococcal A+C Polysaccharide Vaccine
Description: as for outcome 2
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Geometric mean titers were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2)
Number analyzed (Participants) | 304 | 308
Titers
  Serogroup A (pre-vaccination) | 1.71 [1.49 to 1.97] | 1.44 [1.27 to 1.63]
  Serogroup A (post-vaccination) | 203 [178 to 233] | 225 [202 to 250]

6. Secondary Outcome: Geometric Mean Titers of Serogroup C Antibodies Following Vaccination With Either Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine or Lanzhou Institute of Biological Products Meningococcal A+C Polysaccharide Vaccine
Description: as for outcome 3
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination
Population: Geometric mean titers were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2)
Number analyzed (Participants) | 304 | 308
Titers
  Serogroup C (pre-vaccination) | 3.66 [3.27 to 4.10] | 3.64 [3.25 to 4.07]
  Serogroup C (post-vaccination) | 179 [155 to 206] | 191 [167 to 220]

7. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reactions Following Vaccination of Sanofi Pasteur Meningococcal A+C Polysaccharide Vaccine or Lanzhou Institute of Biological Products Meningococcal A+C Polysaccharide Vaccine
Description: Solicited injection site: Pain, Erythema, and Swelling; Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia. Grade 3 injection site: Pain, Incapacitating, unable to perform usual activities; Erythema and Swelling, ≥30 mm. Grade 3 systemic reactions: Fever, temperature >39˚C; Headache, Malaise, and Myalgia, Significant, preventing daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set (SafAS). A Group 2 subject received the wrong vaccine and was included in Full Analysis Set for Group 2 (where classification was per vaccine randomized to) and also Group 1 SafAS (where classification was according to vaccine actually received).
Measure: Number; unit: Participants
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2)
Number analyzed (Participants) | 333 | 332
Participants
  Injection site Pain (N = 331, 331) | 82 | 71 [0 to 0]
  Grade 3 Injection site Pain (N = 331, 331) | 1 | 0 [0 to 0]
  Injection site Erythema (N = 331, 331) | 44 | 32 [0 to 0]
  Grade 3 Injection site Erythema (N = 331, 331) | 1 | 0 [0 to 0]
  Injection site Swelling (N = 331, 331) | 20 | 17 [0 to 0]
  Grade 3 Injection site Swelling (N = 331, 331) | 0 | 1 [0 to 0]
  Fever (N = 330, 330) | 46 | 39 [0 to 0]
  Grade 3 Fever (N = 330, 330) | 1 | 0 [0 to 0]
  Headache (N = 331, 331) | 27 | 20 [0 to 0]
  Grade 3 Headache (N = 331, 331) | 0 | 0 [0 to 0]
  Malaise (N = 331, 331) | 32 | 33 [0 to 0]
  Grade 3 Malaise (N = 331, 331) | 0 | 0 [0 to 0]
  Myalgia (N = 331, 331) | 29 | 42 [0 to 0]
  Grade 3 Myalgia (N = 331, 331) | 0 | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 30 post-vaccination.
Description: A Group 2 subject received the wrong vaccine and was included in Full Analysis Set for Group 2 (classification per vaccine randomized to) and also Group 1 Safety Analysis Set (SafAS, classification according to vaccine actually received). For the solicited injection site and systemic reactions, the total (N) is the number with available data.
Arm/Group | Meningo A+C® (Group 1) | Meng Ling Kang® (Group 2)
Serious Adverse Events (participants affected / at risk) | 2/333 | 1/332
Other Adverse Events (participants affected / at risk) | 82/333 | 71/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meningo A+C® (Group 1) (N=333) | Meng Ling Kang® (Group 2) (N=332)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Meningo A+C® (Group 1) (N=333) | Meng Ling Kang® (Group 2) (N=332)
Nasopharyngitis (Infections and infestations) | 56 (60) | 46 (48)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 29 (32)
Injection site Pain (General disorders) | 82/331 (82) | 71/331 (71)
Injection site Erythema (General disorders) | 44/331 (44) | 32/331 (32)
Injection site Swelling (General disorders) | 20/331 (20) | 17/331 (17)
Fever (General disorders) | 46/330 (46) | 39/330 (39)
Headache (Nervous system disorders) | 27/331 (27) | 20/331 (20)
Malaise (General disorders) | 32/331 (32) | 33/331 (33)
Myalgia (Musculoskeletal and connective tissue disorders) | 29/331 (29) | 42/331 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.